CLINICAL TRIAL: NCT00846807
Title: Observational Cohort Study to Evaluate the Safety and Efficacy of Pradaxa (Dabigatran Etexilate) for the Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Hip Replacement Surgery or Total Knee Replacement Surgery in a Routine Clinical Setting.
Brief Title: Pradaxa (Dabigatran Etexilate 220 mg/q.d. in the General Population After Hip or Knee Replacement Surgery
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.85
Record Dates: First submitted 2009-02-13; First posted 2009-02-19 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Arthroplasty, Replacement; Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients 75 years or younger

SUMMARY:
An observational cohort study on safety and efficacy of the 220 mg dose Pradaxa to generate additional data in predefined sub populations of patients at increased risk of bleeding or VTE

ELIGIBILITY:
Inclusion criteria:

Patients of 18 years of age or above undergoing elective total hip or knee replacement surgery who consent in writing to their participation in this observational study

Exclusion criteria:

All patients who should not be treated with Pradaxa 220 mg according to the European Summary of Product Characteristics (SPC): age of > 75 years, renal impairment (creatinine clearance <50 ml/min), patients with concomitant therapy of amiodarone, elevated liver enzymes > 2 upper limit of normal (ULN) and/or hepatic impairment or liver disease expected to have any impact on survival, anaesthesia with post operative indwelling epidural catheters, hypersensitivity to dabigatran etexilate or to any of the excipients, active clinically significant bleeding, organic lesion at risk of bleeding, spontaneous or pharmacological impairment of haemostasis except for the above included patients groups, concomitant treatment with quinidine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subgroups of the general population
Sampling Method: Non-Probability Sample
Enrollment: 5476 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (112):
- Austria (11):
  - 1160.85.4308 Boehringer Ingelheim Investigational Site, Graz
  - 1160.85.4309 Boehringer Ingelheim Investigational Site, Klagenfurt
  - 1160.85.4303 Boehringer Ingelheim Investigational Site, Linz
  - 1160.85.4304 Boehringer Ingelheim Investigational Site, Linz
  - 1160.85.4305 Boehringer Ingelheim Investigational Site, Saint Johann/Tirol
  - 1160.85.4312 Boehringer Ingelheim Investigational Site, Stolzalpe
  - 1160.85.4301 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.85.4302 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.85.4310 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.85.4311 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.85.4307 Boehringer Ingelheim Investigational Site, Wels
- France (26):
  - 1160.85.3306A Boehringer Ingelheim Investigational Site, Angers
  - 1160.85.3318A Boehringer Ingelheim Investigational Site, Bois Guillaume Cédex
  - 1160.85.3333A Boehringer Ingelheim Investigational Site, Bordeaux
  - 1160.85.3310A Boehringer Ingelheim Investigational Site, Caen
  - 1160.85.3311A Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 1160.85.3315A Boehringer Ingelheim Investigational Site, Créteil
  - 1160.85.3305A Boehringer Ingelheim Investigational Site, Dijon Cédex
  - 1160.85.3304A Boehringer Ingelheim Investigational Site, Illkirch-Graffenstaden
  - 1160.85.3334A Boehringer Ingelheim Investigational Site, Le Havre
  - 1160.85.3324A Boehringer Ingelheim Investigational Site, Les Lilas
  - 1160.85.3309A Boehringer Ingelheim Investigational Site, Lille
  - 1160.85.3307A Boehringer Ingelheim Investigational Site, Lyon
  - 1160.85.3325A Boehringer Ingelheim Investigational Site, Marseille
  - 1160.85.3323A Boehringer Ingelheim Investigational Site, Metz
  - 1160.85.3321A Boehringer Ingelheim Investigational Site, Nantes Cédex 2
  - 1160.85.3301A Boehringer Ingelheim Investigational Site, Paris
  - 1160.85.3302A Boehringer Ingelheim Investigational Site, Paris
  - 1160.85.3303A Boehringer Ingelheim Investigational Site, Paris
  - 1160.85.3320A Boehringer Ingelheim Investigational Site, Paris
  - 1160.85.3308A Boehringer Ingelheim Investigational Site, Pierre-Bénite
  - 1160.85.3322A Boehringer Ingelheim Investigational Site, Poitiers Cédex
  - 1160.85.3319A Boehringer Ingelheim Investigational Site, Saint Etienne Cédex 2
  - 1160.85.3317A Boehringer Ingelheim Investigational Site, Saint-Saulve
  - 1160.85.3314A Boehringer Ingelheim Investigational Site, Toulouse
  - 1160.85.3313A Boehringer Ingelheim Investigational Site, Toulouse Cédex 9
  - 1160.85.3331A Boehringer Ingelheim Investigational Site, Vannes Cédex
- Germany (44):
  - 1160.85.04924 Boehringer Ingelheim Investigational Site, Bad Homburg
  - 1160.85.04926 Boehringer Ingelheim Investigational Site, Bayreuth
  - 1160.85.04903 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.85.04931 Boehringer Ingelheim Investigational Site, Bochum
  - 1160.85.04930 Boehringer Ingelheim Investigational Site, Breitenbrunn
  - 1160.85.04923 Boehringer Ingelheim Investigational Site, Chemnitz
  - 1160.85.04947 Boehringer Ingelheim Investigational Site, Erlangen
  - 1160.85.04945 Boehringer Ingelheim Investigational Site, Fürth
  - 1160.85.04912 Boehringer Ingelheim Investigational Site, Garmische-Partenkirchen
  - 1160.85.04922 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 1160.85.04917 Boehringer Ingelheim Investigational Site, Gelsenkirchen
  - 1160.85.04949 Boehringer Ingelheim Investigational Site, Günzburg
  - 1160.85.04927 Boehringer Ingelheim Investigational Site, Hachenburg
  - 1160.85.04910 Boehringer Ingelheim Investigational Site, Hamburg
  - 1160.85.04906 Boehringer Ingelheim Investigational Site, Hanover
  - 1160.85.04920 Boehringer Ingelheim Investigational Site, Hof
  - 1160.85.04916 Boehringer Ingelheim Investigational Site, Kamp-Linfort
  - 1160.85.04939 Boehringer Ingelheim Investigational Site, Kassel
  - 1160.85.04929 Boehringer Ingelheim Investigational Site, Koblenz
  - 1160.85.04909 Boehringer Ingelheim Investigational Site, Landstuhl
  - 1160.85.04944 Boehringer Ingelheim Investigational Site, Lubin
  - 1160.85.04935 Boehringer Ingelheim Investigational Site, Mainz
  - 1160.85.04902 Boehringer Ingelheim Investigational Site, Marburg
  - 1160.85.04934 Boehringer Ingelheim Investigational Site, Markgröningen
  - 1160.85.04918 Boehringer Ingelheim Investigational Site, Marktheidenfeld
  - 1160.85.04941 Boehringer Ingelheim Investigational Site, Merseburg
  - 1160.85.04952 Boehringer Ingelheim Investigational Site, Minden
  - 1160.85.04943 Boehringer Ingelheim Investigational Site, München
  - 1160.85.04946 Boehringer Ingelheim Investigational Site, München
  - 1160.85.04904 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1160.85.04913 Boehringer Ingelheim Investigational Site, Olsberg
  - 1160.85.04932 Boehringer Ingelheim Investigational Site, Pfortzheim
  - 1160.85.04901 Boehringer Ingelheim Investigational Site, Rosenheim
  - 1160.85.04915 Boehringer Ingelheim Investigational Site, Rostock
  - 1160.85.04928 Boehringer Ingelheim Investigational Site, Rostock
  - 1160.85.04936 Boehringer Ingelheim Investigational Site, Rotenburg/Fulda
  - 1160.85.04905 Boehringer Ingelheim Investigational Site, Schwarzenbruck
  - 1160.85.04914 Boehringer Ingelheim Investigational Site, Sylt
  - 1160.85.04933 Boehringer Ingelheim Investigational Site, Wertheim am Main
  - 1160.85.04921 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 1160.85.04938 Boehringer Ingelheim Investigational Site, Wismar
  - 1160.85.04907 Boehringer Ingelheim Investigational Site, Worms
  - 1160.85.04940 Boehringer Ingelheim Investigational Site, Würzburg
  - 1160.85.04948 Boehringer Ingelheim Investigational Site, Würzburg
- 1160.85.35301 Boehringer Ingelheim Investigational Site, Croom, Ireland
- Italy (10):
  - 1160.85.03911 Boehringer Ingelheim Investigational Site, Bari
  - 1160.85.03905 Boehringer Ingelheim Investigational Site, Florence
  - 1160.85.03904 Boehringer Ingelheim Investigational Site, Genova
  - 1160.85.03906 Boehringer Ingelheim Investigational Site, Jesi (an)
  - 1160.85.03914 Boehringer Ingelheim Investigational Site, Latina
  - 1160.85.03901 Boehringer Ingelheim Investigational Site, Mantova
  - 1160.85.03913 Boehringer Ingelheim Investigational Site, Ome (bs)
  - 1160.85.03907 Boehringer Ingelheim Investigational Site, Roma
  - 1160.85.03909 Boehringer Ingelheim Investigational Site, Torino
  - 1160.85.03910 Boehringer Ingelheim Investigational Site, Vimercate (mi)
- Poland (5):
  - 1160.85.4806 Boehringer Ingelheim Investigational Site, Gmina Świebodzin
  - 1160.85.4805 Boehringer Ingelheim Investigational Site, Kościerzyna
  - 1160.85.4804 Boehringer Ingelheim Investigational Site, Lodz
  - 1160.85.4803 Boehringer Ingelheim Investigational Site, Otwock
  - 1160.85.4802 Boehringer Ingelheim Investigational Site, Piekary Śląskie
- Spain (6):
  - 1160.85.3404 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.85.3406 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.85.3405 Boehringer Ingelheim Investigational Site, Málaga
  - 1160.85.3407 Boehringer Ingelheim Investigational Site, Pamplona
  - 1160.85.3401 Boehringer Ingelheim Investigational Site, Valencia
  - 1160.85.3402 Boehringer Ingelheim Investigational Site, Zaragoza
- Sweden (3):
  - 1160.85.4603 Boehringer Ingelheim Investigational Site, Kungälv
  - 1160.85.4601 Boehringer Ingelheim Investigational Site, Motala
  - 1160.85.4604 Boehringer Ingelheim Investigational Site, Sollefteå
- United Kingdom (6):
  - 1160.85.04405 Boehringer Ingelheim Investigational Site, Basildon
  - 1160.85.04406 Boehringer Ingelheim Investigational Site, Gateshead
  - 1160.85.04402 Boehringer Ingelheim Investigational Site, Halifax
  - 1160.85.04404 Boehringer Ingelheim Investigational Site, London
  - 1160.85.04403 Boehringer Ingelheim Investigational Site, Luton
  - 1160.85.04401 Boehringer Ingelheim Investigational Site, Wigan

REFERENCES:
- [Derived] Rosencher N, Samama CM, Feuring M, Brueckmann M, Kleine E, Clemens A, Frostick S. Dabigatran etexilate for thromboprophylaxis in over 5000 hip or knee replacement patients in a real-world clinical setting. Thromb J. 2016 Apr 1;14:8. doi: 10.1186/s12959-016-0082-4. eCollection 2016. PMID 27042163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 5438 patients enrolled, 5292 were treated. Treated patients are presented.
Pre-assignment Details: Phase IV, open-label, prospective, observational, single-arm study on surgery patients (hip and knee surgery)
Groups:
- All Patients: treated with dabigatran etexilate (Pradaxa), planned dose: 110 mg at the day of surgery, from the day after surgery to last treatment day 220 mg once daily.
Period: Overall Study
Arm/Group | All Patients
Started | 5292 (Entered and treated.)
Completed | 4660 (Completed treatment.)
Not Completed | 632
Not completed — Adverse Event | 270
Not completed — Lost to Follow-up | 94
Not completed — Withdrawal by Subject | 56
Not completed — Non compliant with European label | 7
Not completed — Switch to other anticoagulants | 89
Not completed — No prescription after hospital discharge | 56
Not completed — Other | 60

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 5292
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3061
  Male | 2231

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Major Bleeding Events (MBE) During Treatment Period
Description: Major bleeding events were defined according to the modified McMaster criteria, and were classified by the investigator as Major bleeding event or Any bleeding event. The criteria for MBE's were: fatal; clinically overt associated with loss of haemoglobin >=20g/L in excess of what was expected; clinically overt leading to the transfusion of >=2 units packed cells or whole blood in excess of what was expected; symptomatic retroperitoneal, intracranial, intraocular or intraspinal; requiring treatment cessation; leading to re-operation
Time Frame: From first intake (day of surgery) until 24 hours after last intake (planned: knee replacement: Day 10 after surgery, hip replacement: Day 28-35 after surgery) of Pradaxa
Population: Treated Set (TS) comprises all patients who completed the surgery and received at least 1 dose of dabigatran etexilate.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 5292
Percentage of participants | 0.72 (0.51, 0.98) [0.51 to 0.98]

2. Primary Outcome: Percentage of Patients With Symptomatic Venous Thromboembolic Events (sVTE) and All Cause Mortality
Description: The co-primary efficacy variable sVTE was defined as the composite of documented symptomatic proximal and distal deep vein thrombosis (DVT) and documented symptomatic non-fatal pulmonary embolism (PE).
Time Frame: as for outcome 1
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 5292
Percentage of participants | 1.04 (0.78) [0.78 to 1.35]

3. Secondary Outcome: Percentage of Patients With Major Extra-surgical Site Bleedings
Time Frame: as for outcome 1
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 5292
Percentage of participants | 0.32 ((0.19, 0.51)) [0.19 to 0.51]

4. Secondary Outcome: Volume of Wound Drainage (Post-operative)
Description: Total volume of wound drainage is calculated as sum of volume drainage from end of surgery until first dose of Pradaxa plus volume drainage from first dose of Pradaxa and onwards.
Time Frame: From end of surgery (before first dosing) until 24 hours after last intake (planned: knee replacement: Day 10 after surgery, hip replacement: Day 28-35 after surgery) of Pradaxa
Population: TS
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | All Patients
Number analyzed (Participants) | 4228
ml | 704.5 (418.0)

5. Secondary Outcome: Percentage of Patients With Single Components of Composite of sVTE and All-cause Mortality
Time Frame: as for outcome 1
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 5292
Percentage of participants
  Documented symptomatic proximal DVT | 0.17 ((0.08, 0.32)) [0.08 to 0.32]
  Documented symptomatic distal DVT | 0.87 ((0.64, 1.16)) [0.64 to 1.16]
  Documented symptomatic non-fatal PE | 0.09 ((0.03, 0.22)) [0.03 to 0.22]
  All-cause mortality | 0.06 ((0.01, 0,17)) [0.01 to 0.17]

ADVERSE EVENTS:
Time Frame: From first intake (day of surgery) until 24 hours after last intake (planned: knee replacement: Day 10 after surgery, hip replacement: Day 28-35 after surgery) of Pradaxa
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 135/5292
Other Adverse Events (participants affected / at risk) | 0/5292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=5292)
Pneumonia (Infections and infestations) | 4
Postoperative wound infection (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 2
Peritoneal infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Coagulation factor deficiency (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Allergy to metals (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Monoparesis (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Vitreous detachment (Eye disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Myocardial ischaemia (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Deep vein thrombosis (Vascular disorders) | 9
Haematoma (Vascular disorders) | 7
Haemorrhage (Vascular disorders) | 5
Thrombophlebitis superficial (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Scar (Skin and subcutaneous tissue disorders) | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 4
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint lock (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Device dislocation (General disorders) | 8
Drug ineffective (General disorders) | 8
Oedema peripheral (General disorders) | 4
Adverse drug reaction (General disorders) | 1
Asthenia (General disorders) | 1
Death (General disorders) | 2
Pyrexia (General disorders) | 2
Blood glucose increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Fat embolism (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 6
Joint dislocation (Injury, poisoning and procedural complications) | 3
Operative haemorrhage (Injury, poisoning and procedural complications) | 6
Wound dehiscence (Injury, poisoning and procedural complications) | 6
Wound secretion (Injury, poisoning and procedural complications) | 5
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Joint sprain (Injury, poisoning and procedural complications) | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1
Rehabilitation therapy (Surgical and medical procedures) | 1
Immobilisation prolonged (Social circumstances) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.